CLINICAL TRIAL: NCT06424236
Title: A Phase II/III Multicenter Randomized, Double-Blind, Placebo-Controlled Platform Trial of Potential Disease Modifying Therapies Utilizing Biomarker, Cognitive, and Clinical Endpoints in Dominantly Inherited Alzheimer's Disease
Brief Title: Dominantly Inherited Alzheimer Network Trial: An Opportunity to Prevent Dementia: A Study of Potential Disease Modifying Treatments in Individuals at Risk for or With a Type of Early Onset Alzheimer's Disease Caused by a Genetic Mutation
Acronym: DIAN-TU
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DIAN-TU announced the discontinuation of the DIAN-TU-001 OLE based on the status of the drug program and findings from an interim efficacy analysis and.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Hoffmann-La Roche (Industry); Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAN-TU-001 (Gant OLE); The Alzheimer's Association (Other Grant/Funding Number: DIAN TTU-12-243040); U01AG042791 (NIH); 2013-000307-17 (EudraCT Number); R01AG046179 (NIH); REec-2014-0817 (Registry Identifier: Spanish Clinical Studies Registry); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU Tau-15-347219); GHR Foundation (Other Grant/Funding Number: File 4401); Alzheimer's Association (Other: HDE 18S84914); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU NG-16-434362); R56AG053267 (NIH); U01AG059798 (NIH); R01AG053267 (NIH)
Record Dates: First submitted 2024-04-16; First posted 2024-05-22 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — gantenerumab

STUDY DESIGN:
Masking Description: Arm is Open-label as noted in the arm description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gantenerumab Open Label Extension (Experimental): Gantenerumab: Subcutaneously every 4 weeks, at escalating doses; at target, dosing was every 2 weeks
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Open-label administered Subcutaneously every 4 weeks, at escalating doses; at target, dosing was every 2 weeks
  Other Names: RO4909832

SUMMARY:
The purpose of this study is to assess the safety, tolerability, biomarker, cognitive and clinical efficacy of investigational products in participants with an Alzheimer's disease-causing mutation by determining if treatment with the study drug slows the rate of progression of cognitive/clinical impairment or improves disease-related biomarkers.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is defined by the presence of abnormal accumulations of amyloid protein (plaques) and tau protein (tangles) in the brain. The double-blind arm of DIAN-TU-001 Master protocol (NCT01760005) tested whether gantenerumab provided a clinical benefit by slowing the onset or the worsening of the disease. A clinical benefit was not observed in the double-blind part of the DIAN-TU-001 study. However, gantenerumab was associated with improvements in measures of amyloid and tau and an improvement in an overall measure of neurodegeneration (when nerve cells in the brain lose function over time). It is not known whether these changes may provide future clinical benefits. Based on this information, an exploratory Open Label Extension (OLE) will further study the effect of gantenerumab on these Alzheimer-related proteins and their relationship to disease progression.

After this final evaluation of study treatment with gantenerumab used in the gantenerumab / solanezumab double-blind arm of the Master protocol (NCT01760005), eligible participants from the placebo, solanezumab, and gantenerumab treatment groups in double-blind period were invited to participate in an OLE period to receive active gantenerumab study treatment as part of the DIAN-TU-001 Master protocol. The OLE period of the study planned to provide study treatment with gantenerumab for up to 3 years (36 months).

This study collected brain scans, blood, and spinal fluid tests (also called biomarkers), as well as safety, clinical and cognitive testing. The goal is to determine if gantenerumab has favorable effects on these tests to determine if and how much treatment may prevent or delay the symptoms of AD.

Update:

Based on the results of the completed studies of gantenerumab in sporadic AD in late 2022, it was decided to determine if dominantly inherited Alzheimer's disease (DIAD) participants in the DIAN-TU-001 OLE study were substantially clinically benefiting from gantenerumab high-dose treatment before the trial reached completion as the Gant program was being stopped.

An interim efficacy analysis of the DIAN-TU-001 OLE was performed to:

1. determine if gantenerumab OLE treatment and/or long-term treatment results in clinical benefit and determine the extent of amyloid removal compared to the double-blind period.
2. determine the potential effects of gantenerumab on clinical and cognitive measures to support decision-making regarding next steps for the DIAN-TU-001 OLE.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-80 years of age
* Individuals who know they have an Alzheimer's disease-causing mutation
* Individuals who have participated in the double-blind period
* In the opinion of the investigator and sponsor, treatment is not contraindicated for safety
* Capable of receiving drug and appropriate clinical safety assessment
* Able to undergo Magnetic Resonance Imaging (MRI), Lumbar Puncture (LP), Positron Emission Tomography (PET), and complete all study related testing and evaluations.
* For women of childbearing potential, if partner is not sterilized, subject must agree to use effective contraceptive measures (hormonal contraception, intra-uterine device, sexual abstinence, barrier method with spermicide).
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.
* Has a Study Partner who in the investigator's judgment is able to provide accurate information as to the subject's cognitive and functional abilities, who agrees to provide information at the study visits which require informant input for scale completion.

Exclusion Criteria:

* History or presence of brain MRI scans indicative of any other significant abnormality
* Alcohol or drug dependence currently or within the past 1 year
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would preclude MRI scan.
* History or presence of clinically significant cardiovascular disease, hepatic/renal disorders, infectious disease or immune disorder, or metabolic/endocrine disorders
* Anticoagulants except low dose (≤ 325 mg) aspirin.
* Have been exposed to a monoclonal antibody targeting beta amyloid peptide within the past six months.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
* Positive urine or serum pregnancy test or plans or desires to become pregnant during the course of the trial.
* Subjects unable to complete all study related testing, including implanted metal that cannot be removed for MRI scanning, required anticoagulation and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Bateman, MD, Study Director — Washington University School of Medicine
Locations (17):
- United States (8):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - University of Washington, Seattle, Washington
- Australia (3):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
  - The McCuster Foundation of Alzheimer's Disease Research, Nedlands, Western Australia
- France (3):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].

REFERENCES:
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Farlow M, Arnold SE, van Dyck CH, Aisen PS, Snider BJ, Porsteinsson AP, Friedrich S, Dean RA, Gonzales C, Sethuraman G, DeMattos RB, Mohs R, Paul SM, Siemers ER. Safety and biomarker effects of solanezumab in patients with Alzheimer's disease. Alzheimers Dement. 2012 Jul;8(4):261-71. doi: 10.1016/j.jalz.2011.09.224. Epub 2012 Jun 5. PMID 22672770
- [Background] Bateman RJ, Benzinger TL, Berry S, Clifford DB, Duggan C, Fagan AM, Fanning K, Farlow MR, Hassenstab J, McDade EM, Mills S, Paumier K, Quintana M, Salloway SP, Santacruz A, Schneider LS, Wang G, Xiong C; DIAN-TU Pharma Consortium for the Dominantly Inherited Alzheimer Network. The DIAN-TU Next Generation Alzheimer's prevention trial: Adaptive design and disease progression model. Alzheimers Dement. 2017 Jan;13(1):8-19. doi: 10.1016/j.jalz.2016.07.005. Epub 2016 Aug 29. PMID 27583651
- [Background] Mills SM, Mallmann J, Santacruz AM, Fuqua A, Carril M, Aisen PS, Althage MC, Belyew S, Benzinger TL, Brooks WS, Buckles VD, Cairns NJ, Clifford D, Danek A, Fagan AM, Farlow M, Fox N, Ghetti B, Goate AM, Heinrichs D, Hornbeck R, Jack C, Jucker M, Klunk WE, Marcus DS, Martins RN, Masters CM, Mayeux R, McDade E, Morris JC, Oliver A, Ringman JM, Rossor MN, Salloway S, Schofield PR, Snider J, Snyder P, Sperling RA, Stewart C, Thomas RG, Xiong C, Bateman RJ. Preclinical trials in autosomal dominant AD: implementation of the DIAN-TU trial. Rev Neurol (Paris). 2013 Oct;169(10):737-43. doi: 10.1016/j.neurol.2013.07.017. Epub 2013 Sep 6. PMID 24016464
- [Background] Wang G, Berry S, Xiong C, Hassenstab J, Quintana M, McDade EM, Delmar P, Vestrucci M, Sethuraman G, Bateman RJ; Dominantly Inherited Alzheimer Network Trials Unit. A novel cognitive disease progression model for clinical trials in autosomal-dominant Alzheimer's disease. Stat Med. 2018 Sep 20;37(21):3047-3055. doi: 10.1002/sim.7811. Epub 2018 May 14. PMID 29761523
- [Background] Weninger S, Carrillo MC, Dunn B, Aisen PS, Bateman RJ, Kotz JD, Langbaum JB, Mills SL, Reiman EM, Sperling R, Santacruz AM, Tariot PN, Welsh-Bohmer KA. Collaboration for Alzheimer's Prevention: Principles to guide data and sample sharing in preclinical Alzheimer's disease trials. Alzheimers Dement. 2016 May;12(5):631-2. doi: 10.1016/j.jalz.2016.04.001. No abstract available. PMID 27157073
- [Background] Grill JD, Bateman RJ, Buckles V, Oliver A, Morris JC, Masters CL, Klunk WE, Ringman JM; Dominantly Inherited Alzheimer's Network. A survey of attitudes toward clinical trials and genetic disclosure in autosomal dominant Alzheimer's disease. Alzheimers Res Ther. 2015 Jul 22;7(1):50. doi: 10.1186/s13195-015-0135-0. eCollection 2015. PMID 26203303
- [Background] McDade E, Bateman RJ. Stop Alzheimer's before it starts. Nature. 2017 Jul 12;547(7662):153-155. doi: 10.1038/547153a. No abstract available. PMID 28703214
- [Background] McDade E, Wang G, Gordon BA, Hassenstab J, Benzinger TLS, Buckles V, Fagan AM, Holtzman DM, Cairns NJ, Goate AM, Marcus DS, Morris JC, Paumier K, Xiong C, Allegri R, Berman SB, Klunk W, Noble J, Ringman J, Ghetti B, Farlow M, Sperling RA, Chhatwal J, Salloway S, Graff-Radford NR, Schofield PR, Masters C, Rossor MN, Fox NC, Levin J, Jucker M, Bateman RJ; Dominantly Inherited Alzheimer Network. Longitudinal cognitive and biomarker changes in dominantly inherited Alzheimer disease. Neurology. 2018 Oct 2;91(14):e1295-e1306. doi: 10.1212/WNL.0000000000006277. Epub 2018 Sep 14. PMID 30217935
- [Background] Ryman DC, Acosta-Baena N, Aisen PS, Bird T, Danek A, Fox NC, Goate A, Frommelt P, Ghetti B, Langbaum JB, Lopera F, Martins R, Masters CL, Mayeux RP, McDade E, Moreno S, Reiman EM, Ringman JM, Salloway S, Schofield PR, Sperling R, Tariot PN, Xiong C, Morris JC, Bateman RJ; Dominantly Inherited Alzheimer Network. Symptom onset in autosomal dominant Alzheimer disease: a systematic review and meta-analysis. Neurology. 2014 Jul 15;83(3):253-60. doi: 10.1212/WNL.0000000000000596. Epub 2014 Jun 13. PMID 24928124
- [Background] Weng H, Bateman R, Morris JC, Xiong C. Validity and power of minimization algorithm in longitudinal analysis of clinical trials. Biostat Epidemiol. 2017;1(1):59-77. doi: 10.1080/24709360.2017.1331822. Epub 2017 Jun 13. PMID 29250611
- [Result] Bateman, Randall J., Yan Li, Eric McDade, Jorge J. Llibre Guerra, David Clifford, Alireza Atri, Susan Mills, et al. "Amyloid Reduction and Dementia Progression in Dominantly Inherited Alzheimer's Disease after Long-Term Gantenerumab Treatment: Results from the Dian-Tu Trial." SSRN Scholarly Paper. Rochester, NY, July 26, 2024. https://doi.org/10.2139/ssrn.4906344.
- [Derived] Bateman RJ, Li Y, McDade EM, Llibre-Guerra JJ, Clifford DB, Atri A, Mills SL, Santacruz AM, Wang G, Supnet C, Benzinger TLS, Gordon BA, Ibanez L, Klein G, Baudler M, Doody RS, Delmar P, Kerchner GA, Bittner T, Wojtowicz J, Bonni A, Fontoura P, Hofmann C, Kulic L, Hassenstab J, Aschenbrenner AJ, Perrin RJ, Cruchaga C, Renton AE, Xiong C, Goate AA, Morris JC, Holtzman DM, Snider BJ, Mummery C, Brooks WS, Wallon D, Berman SB, Roberson E, Masters CL, Galasko DR, Jayadev S, Sanchez-Valle R, Pariente J, Kinsella J, van Dyck CH, Gauthier S, Hsiung GR, Masellis M, Dubois B, Honig LS, Jack CR, Daniels A, Aguillon D, Allegri R, Chhatwal J, Day G, Fox NC, Huey E, Ikeuchi T, Jucker M, Lee JH, Levey AI, Levin J, Lopera F, Roh J, Rosa-Neto P, Schofield PR; Dominantly Inherited Alzheimer's Disease-Trials Unit. Safety and efficacy of long-term gantenerumab treatment in dominantly inherited Alzheimer's disease: an open-label extension of the phase 2/3 multicentre, randomised, double-blind, placebo-controlled platform DIAN-TU trial. Lancet Neurol. 2025 Apr;24(4):316-330. doi: 10.1016/S1474-4422(25)00024-9. PMID 40120616
- [Derived] Bateman RJ, Li Y, McDade EM, Llibre-Guerra JJ, Clifford DB, Atri A, Mills SL, Santacruz AM, Wang G, Supnet C, Benzinger TLS, Gordon BA, Ibanez L, Klein G, Baudler M, Doody RS, Delmar P, Kerchner GA, Bittner T, Wojtowicz J, Bonni A, Fontoura P, Hofmann C, Kulic L, Hassenstab J, Aschenbrenner AJ, Perrin RJ, Cruchaga C, Renton AE, Xiong C, Goate AA, Morris JC, Holtzman DM, Snider BJ, Mummery C, Brooks WS, Wallon D, Berman SB, Roberson E, Masters CL, Galasko DR, Jayadev S, Sanchez-Valle R, Pariente J, Kinsella J, van Dyck CH, Gauthier S, Robin Hsiung GY, Masellis M, Dubois B, Honig LS, Jack CR, Daniels A, Aguillon D, Allegri R, Chhatwal J, Day G, Fox N, Huey E, Ikeuchi T, Jucker M, Lee JH, Levey AI, Levin J, Lopera F, Roh J, Rosa-Neto P, Schofield PR; Dominantly Inherited Alzheimer's Disease-Trials Unit. Safety and efficacy of long-term gantenerumab treatment in dominantly inherited Alzheimer's disease: an open label extension of the phase 2/3 multicentre, randomised, double-blind, placebo-controlled platform DIAN-TU Trial. medRxiv [Preprint]. 2025 Jan 29:2024.10.29.24316289. doi: 10.1101/2024.10.29.24316289. PMID 39974075
- See also: Expanded registry — http://www.dianexr.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a open-label period of the trial following a Phase II/III double-blind, placebo-controlled study conducted in participants with, or at risk for, dominantly inherited Alzheimer's disease at 17 sites in the United States, Canada, Australia and Europe between 03 June 2020 and 13 November 2023.
Pre-assignment Details: All eligible participants from DIAN-TU-001 trial sites were offered the opportunity to receive gantenerumab for up to 3 years in an open-label extension (OLE). A total of 74 participants were enrolled in the OLE period of which, 1 participant was screen failure.
Groups:
- Double-blind Placebo - OLE Gantenerumab: Eligible participants from placebo treatment group in double-blind period entered OLE period to receive gantenerumab up to 1500 milligram (mg) subcutaneous (SC) infusion every 2 weeks (Q2W) for 3 years.
- Double-blind Solanezumab - OLE Gantenerumab: Eligible participants from solanezumab treatment group in double-blind period entered OLE period to receive gantenerumab up to 1500 mg SC infusion Q2W for 3 years.
- Double-blind Gantenerumab - OLE Gantenerumab: Eligible participants from gantenerumab treatment group in double-blind period entered OLE period to continue to receive gantenerumab up to 1500 mg SC infusion Q2W for 3 years.
Period: Overall Study
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Started | 18 | 27 | 28
Completed | 4 | 2 | 7
Not Completed | 14 | 25 | 21
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 11 | 20 | 16
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who received at least 1 dose of study drug in the gantenerumab OLE period.
Groups:
- Double-blind Placebo - OLE Gantenerumab: Eligible participants from placebo treatment group in double-blind period entered OLE period to receive gantenerumab up to 1500 mg SC infusion Q2W for 3 years.
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab | Total
Number analyzed (Participants) | 18 | 27 | 28 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (9.62) | 47.0 (8.60) | 50.3 (7.97) | 48.9 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 13 | 38
  Male | 7 | 13 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 4 | 9
  Not Hispanic or Latino | 14 | 26 | 24 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 26 | 26 | 66
  Black or African American | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Pacific Islanders | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Other | 4 | 1 | 1 | 6
  Unknown | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Composite [11C] Pittsburgh Compound B (PiB)-Positron Emission Tomography (PET) Composite Standardized Uptake Value Ratio (C-SUVR) at Weeks 52, 104 and 156
Description: The composite PiB partial volume corrected C-SUVR was used as the biomarker endpoint for amyloid deposition using PET. The C-SUVR of precuneus, caudate, gyrus rectus, occipital cortex, parietal cortex, prefrontal cortex, and temporal cortex of brain regions was analyzed. Higher ratio indicate worse disease stage. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: The OLE gantenerumab modified intent-to-treat (mITT) analysis set included all participants in the OLE who met mITT criteria using OLE baseline as the baseline reference point. Only participants analyzed at baseline and specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 12 | 20 | 20
ratio
  Week 52: number analyzed (Participants) | 12 | 18 | 14
  Week 52 | -0.1382 (0.22606) | -0.3318 (0.40538) | 0.1201 (0.15142)
  Week 104: number analyzed (Participants) | 10 | 20 | 20
  Week 104 | -0.4843 (0.55217) | -0.7026 (0.63641) | -0.1880 (0.26639)
  Week 156: number analyzed (Participants) | 6 | 9 | 10
  Week 156 | -0.7660 (0.64108) | -1.1761 (0.96831) | -0.2748 (0.41027)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 52: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline Composite [11C] PiB-PET SUVR score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Superiority; p = 0.0117, Mixed Model for Repeated Measures (MMRM); Least square (LS) mean = -0.1166, 95% CI 2-sided [-0.2060 to -0.0272], Standard Deviation 0.29505
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 104: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline Composite [11C] PiB-PET SUVR score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = -0.4648, 95% CI 2-sided [-0.5971 to -0.3326], Standard Deviation 0.46591
Statistical Analysis 3: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 156: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline Composite [11C] PiB-PET SUVR score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = -0.7062, 95% CI 2-sided [-0.8821 to -0.5303], Standard Deviation 0.43787

2. Secondary Outcome: Change From Baseline in Clinical Dementia Rating (CDR) - Sum of Boxes Score at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by CDR - sum of boxes. The CDR-SB score is considered a more detailed quantitative general index of cognition and function than the global CDR score. The CDR - sum of boxes is the sum score of 6 domains of cognitive function (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care), with the score of each domain ranging from 0 (no impairment) to 3 (severe impairment). The total score ranges from 0 (no impairment) to 18 (severe impairment). Higher score indicates worse performance. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: The OLE gantenerumab mITT analysis set included all participants in the OLE who met mITT criteria using OLE baseline as the baseline reference point. Only participants analyzed at baseline and specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 23 | 22
score on a scale
  Week 52 | 1.12 (2.147) | 0.91 (1.497) | 0.09 (0.666)
  Week 104: number analyzed (Participants) | 15 | 21 | 22
  Week 104 | 1.47 (2.191) | 1.31 (2.507) | 0.50 (1.504)
  Week 156: number analyzed (Participants) | 10 | 10 | 14
  Week 156 | 2.15 (3.504) | 0.40 (0.907) | 1.14 (2.405)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; The time to recurrent progression in CDR - sum of boxes. Baseline Asymptomatic Participants: Estimate and confidence interval was based on the Cox proportional hazards regression model including treatment and baseline estimated years to symptom onset as fixed effects. The OLE gantenerumab mITT analysis set included all participants in the OLE who met mITT criteria using OLE baseline as the baseline reference point; Test type: Superiority — Recurrent progression was defined as any progression which was either the first increase in CDR-SB above baseline or any progression above the highest preceding post-baseline value identified as a progression, where progression above the preceding value must be observed at 2 consecutive measurements unless the progression occurs at the last measurement; p = 0.4535, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.64 to 2.70]
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; The time to recurrent progression in CDR - sum of boxes. Baseline Symptomatic Participants: Estimate and confidence interval was based on the Cox proportional hazards regression model including treatment and baseline estimated years to symptom onset as fixed effects. The OLE gantenerumab mITT analysis set included all participants in the OLE who met mITT criteria using OLE baseline as the baseline reference point; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.4848, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.74 to 1.86]

3. Secondary Outcome: Change From Baseline in Clinical Dementia Rating - Global Score at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by CDR - global score. The score ranges from 0 (minimum) to 3 (maximum). Higher score indicates worse performance. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 23 | 22
score on a scale
  Week 52 | 0.12 (0.281) | 0.17 (0.324) | 0.02 (0.188)
  Week 104: number analyzed (Participants) | 15 | 21 | 22
  Week 104 | 0.17 (0.309) | 0.21 (0.514) | 0.09 (0.366)
  Week 156: number analyzed (Participants) | 10 | 10 | 14
  Week 156 | 0.25 (0.425) | 0.10 (0.211) | 0.18 (0.421)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Time to first progression in CDR-Global score. Baseline Asymptomatic Participants: Estimate and confidence interval was based on Cox proportional hazards regression model including treatment and baseline estimated years to symptom onset as fixed effects. Time to first progression was defined as time from baseline to first visit where CDR-Global Score was greater than baseline value, where progression must be observed at 2 consecutive measurements unless progression occurs at last measurement; Test type: Other; p = 0.8855, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.33 to 2.58]
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Time to first progression in CDR-Global score. Baseline Symptomatic Participants: Estimate and confidence interval was based on Cox proportional hazards regression model including treatment and baseline estimated years to symptom onset as fixed effects. Time to first progression was defined as time from baseline to first visit where CDR-Global Score was greater than baseline value, where progression must be observed at 2 consecutive measurements unless progression occurs at last measurement; Test type: Other; p = 0.4497, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.30 to 1.69]

4. Secondary Outcome: Change From Baseline in Functional Assessment Scale (FAS) at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by FAS. This scale measured instrumental activities of daily living such as preparing balanced meals and managing personal finances. The intent of the FAS was to assess change in an individual's functional activities, relative to previously attained abilities, that were caused by cognitive dysfunction. The score ranges from 0 (minimum) to 30 (maximum). Higher score indicates worse performance. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 15 | 22 | 23
score on a scale
  Week 52 | 1.7555 (3.25466) | 1.1060 (2.80472) | 0.4348 (1.67403)
  Week 104: number analyzed (Participants) | 14 | 21 | 23
  Week 104 | 3.1885 (5.48051) | 1.9524 (3.85326) | 0.8889 (2.71006)
  Week 156: number analyzed (Participants) | 9 | 8 | 13
  Week 156 | 2.1944 (3.37680) | 1.0000 (2.39046) | 1.6154 (3.37980)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Baseline Asymptomatic Participants: The statistical model included time since baseline (years), treatment arm, an interaction between treatment and time. Time was considered as continuous. Random intercepts and slopes for each participant was included as random effects with compound symmetry covariance matrix; Test type: Superiority; p = 0.760, Linear Mixed Effects Model; LS mean = -0.06, 95% CI 2-sided [-0.46 to 0.33], Standard Error of Mean 0.200 — Estimated value is the difference in the rate of change between the treatment group and control group
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Baseline Symptomatic Participants: The statistical model included time since baseline (years), treatment arm, an interaction between treatment and time. Time was considered as continuous. Random intercepts and slopes for each participant was included as random effects with an unstructured covariance matrix; Test type: Other; p = 0.093, Linear Mixed Effects Model; LS mean = -1.21, 95% CI 2-sided [-2.63 to 0.20], Standard Error of Mean 0.715 — Estimated value is the difference in the rate of change between the treatment group and control group

5. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) at Weeks 24, 52, 76, 104, 128 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by MMSE. The MMSE is a brief, quantitative measure of cognitive status in adults used to screen for cognitive impairment. The score ranges from 0 (minimum) to 30 (maximum). Lower score indicates worse performance. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 24, 52, 76, 104, 128 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 24 | 24
score on a scale
  Week 24: number analyzed (Participants) | 17 | 22 | 24
  Week 24 | -0.6 (2.40) | -0.5 (3.00) | -0.1 (1.23)
  Week 52 | -1.2 (2.74) | -1.0 (2.47) | -0.9 (2.35)
  Week 76: number analyzed (Participants) | 16 | 22 | 23
  Week 76 | -2.1 (3.70) | -0.8 (3.51) | -0.9 (2.89)
  Week 104: number analyzed (Participants) | 15 | 21 | 24
  Week 104 | -3.1 (5.13) | -1.5 (4.73) | -1.2 (3.53)
  Week 128: number analyzed (Participants) | 11 | 14 | 19
  Week 128 | -3.3 (5.50) | -0.2 (1.93) | -2.1 (4.71)
  Week 156: number analyzed (Participants) | 8 | 6 | 12
  Week 156 | -3.8 (7.61) | 1.2 (1.33) | -1.4 (3.92)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Baseline Asymptomatic Participants: The statistical model included time since baseline (years), treatment arm, an interaction between treatment and time. Time was considered as continuous. Random intercepts and slopes for each participant was included as random effects with an unstructured covariance matrix; Test type: Other; p = 0.989, Linear Mixed Effects Model; LS mean = 0.00, 95% CI 2-sided [-0.43 to 0.44], Standard Error of Mean 0.220 — Estimated value is the difference in the rate of change between the treatment group and control group
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.714, Linear Mixed Effects Model; LS mean = 0.20, 95% CI 2-sided [-0.86 to 1.25], Standard Error of Mean 0.533 — Estimated value is the difference in the rate of change between the treatment group and control group

6. Secondary Outcome: Change From Baseline in Tau Positron Emission Tomography Binding Partial Volume Corrected Standardized Uptake Value Ratio (Tau PET SUVR) at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by Tau PET SUVR. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 12 | 14 | 16
ratio
  Week 52: number analyzed (Participants) | 11 | 13 | 13
  Week 52 | 0.09032 (0.337016) | -0.11554 (0.537111) | 0.12246 (0.202397)
  Week 104 | 0.29471 (0.658922) | 0.19329 (0.811715) | 0.26572 (0.314147)
  Week 156: number analyzed (Participants) | 3 | 4 | 8
  Week 156 | 0.38857 (0.475259) | -0.02390 (0.860703) | 0.21449 (0.281091)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.738, Linear Mixed Effects Model; LS mean = -0.03, 95% CI 2-sided [-0.18 to 0.13], Standard Error of Mean 0.077 — Estimated value is the difference in the rate of change between the treatment group and control group
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.395, Linear Mixed Effects Model; LS mean = 0.19, 95% CI 2-sided [-0.28 to 0.66], Standard Error of Mean 0.222 — Estimated value is the difference in the rate of change between the treatment group and control group

7. Secondary Outcome: Change From Baseline in Phosphorylated Tau (pTau)-181 in Cerebrospinal Fluid (CSF) at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by CSF pTau-181. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 20 | 21
picogram per milliliter (pg/mL)
  Week 52: number analyzed (Participants) | 17 | 19 | 21
  Week 52 | -3.29012 (3.301052) | -2.95397 (3.225444) | -0.28807 (1.740518)
  Week 104: number analyzed (Participants) | 15 | 20 | 21
  Week 104 | -7.15305 (5.152265) | -6.03388 (4.745042) | -1.19673 (2.262092)
  Week 156: number analyzed (Participants) | 9 | 9 | 13
  Week 156 | -8.13416 (5.861080) | -6.83542 (3.548298) | -1.48436 (2.746503)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 56: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF pTau181 as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = -2.1760, 95% CI 2-sided [-2.9469 to -1.4051], Standard Deviation 2.89551
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab; Week 104: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF pTau181 as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = -4.8434, 95% CI 2-sided [-5.8609 to -3.8260], Standard Deviation 3.78771
Statistical Analysis 3: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 156: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF pTau181 as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = -5.7620, 95% CI 2-sided [-6.9679 to -4.5561], Standard Deviation 3.31129

8. Secondary Outcome: Change From Baseline in Neurofilament Light Chain (NfL) in Cerebrospinal Fluid at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by CSF NfL. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 16 | 20 | 21
pg/mL
  Week 52: number analyzed (Participants) | 16 | 19 | 21
  Week 52 | 176.01 (223.432) | 283.97 (255.009) | 106.09 (252.328)
  Week 104: number analyzed (Participants) | 15 | 20 | 20
  Week 104 | 263.74 (268.343) | 351.02 (312.203) | 257.12 (255.528)
  Week 156: number analyzed (Participants) | 9 | 8 | 13
  Week 156 | 233.30 (186.805) | 609.45 (549.253) | 402.20 (536.504)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Baseline Asymptomatic Participants: The statistical model included time since baseline (years), treatment arm, an interaction between treatment and time. Time was considered as continuous. Random intercepts and slopes for each participant was included as random effects with variance components covariance matrix; Test type: Other; p = 0.055, Linear Mixed Effects Model; LS mean = 0.04, 95% CI 2-sided [0.00 to 0.09], Standard Error of Mean 0.022 — Estimated value is the difference in the rate of change between the treatment group and control group
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.188, Linear Mixed Effects Model; LS mean = 0.04, 95% CI 2-sided [-0.02 to 0.11], Standard Error of Mean 0.034 — Estimated value is the difference in the rate of change between the treatment group and control group

9. Secondary Outcome: Change From Baseline in Amyloid Beta1-42/40 Ratio in Cerebrospinal Fluid at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by CSF Amyloid Beta1-42/40. Baseline was defined as the last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 20 | 21
ratio
  Week 52: number analyzed (Participants) | 17 | 19 | 21
  Week 52 | 0.00669 (0.015517) | 0.01217 (0.013657) | -0.00060 (0.008280)
  Week 104: number analyzed (Participants) | 15 | 20 | 20
  Week 104 | 0.02961 (0.022677) | 0.03588 (0.025329) | 0.00571 (0.010013)
  Week 156: number analyzed (Participants) | 9 | 9 | 12
  Week 156 | 0.04400 (0.024807) | 0.05304 (0.037927) | 0.01182 (0.022581)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 52: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF Amyloid Beta1-42/40 score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p = 0.0001, MMRM; LS mean = 0.0067, 95% CI 2-sided [0.0034 to 0.0100], Standard Deviation 0.01240
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 104: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF Amyloid Beta1-42/40 score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = 0.0251, 95% CI 2-sided [0.0189 to 0.0312], Standard Deviation 0.02262
Statistical Analysis 3: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; Week 156: Treatment group and visit were treated as categorical fixed effects factors and OLE baseline CSF Amyloid Beta1-42/40 score as continuous. An unstructured correlation pattern was used to estimate the variance-covariance of the within participant repeated measures. The Kenward-Roger method was used to estimate the denominator degrees of freedom; Test type: Other; p < 0.0001, MMRM; LS mean = 0.0357, 95% CI 2-sided [0.0266 to 0.0447], Standard Deviation 0.02467

10. Secondary Outcome: Change From Baseline in DIAN-TU Open Label Extension Cognitive Composite Score at Weeks 52, 104 and 156
Description: The efficacy of gantenerumab in reducing disease progression was assessed by DIAN-TU OLE Cognitive Composite. The cognitive composite was calculated based on the below 4 components,
  1. The wechsler adult intelligence scale-revised digit span (backward recall). Score ranges from 0 (minimum) to 7 (maximum).
  2. The category fluency (animals) value. Score ranges from 0 to unlimited.
  3. The wechsler adult intelligence scale digit symbol substitution test. Score ranges from 0 (minimum) to 93 (maximum).
  4. The MMSE. Score ranges from 0 (minimum) to 30 (maximum).
  Lower scores of each component indicate worse performance. The cognitive composite is a normalized z score and has score range - 4.11 to unlimited as one of the components has score range 0 to unlimited. Lower score indicates worse performance. Baseline was defined as last non-missing measurement prior to OLE study drug administration.
Time Frame: Baseline (Day 1) and Weeks 52, 104 and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
Number analyzed (Participants) | 17 | 22 | 23
score on a scale
  Week 52 | -0.2281 (0.44682) | -0.1462 (0.37510) | -0.1336 (0.26523)
  Week 104: number analyzed (Participants) | 15 | 21 | 23
  Week 104 | -0.5535 (0.82376) | -0.2373 (0.49333) | -0.2493 (0.48045)
  Week 156: number analyzed (Participants) | 9 | 8 | 12
  Week 156 | -0.3309 (0.60877) | -0.2738 (0.49439) | -0.1327 (0.31666)
Statistical Analysis 1: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.644, Linear Mixed Effects Model; LS mean = 0.04, 95% CI 2-sided [-0.12 to 0.20], Standard Error of Mean 0.081 — Estimated value is the difference in the rate of change between the treatment group and control group
Statistical Analysis 2: Comparison: Double-blind Placebo - OLE Gantenerumab vs Double-blind Solanezumab - OLE Gantenerumab vs Double-blind Gantenerumab - OLE Gantenerumab; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.745, Linear Mixed Effects Model; LS mean = 0.04, 95% CI 2-sided [-0.18 to 0.26], Standard Error of Mean 0.111 — Estimated value is the difference in the rate of change between the treatment group and control group

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from the first dose administration of the OLE study drug (Day 1) up to early termination of study, approximately 156 weeks.
Description: The safety analysis population included all participants who received at least 1 dose of study drug in the gantenerumab OLE period. Only TEAEs that started or worsened in severity on or after first dose of study drug are reported. TEAEs occurred prior to first dose of study drug are not reported as it was pre-specified to report only TEAEs that started or worsened in severity on or after first dose of study drug.
Arm/Group | Double-blind Placebo - OLE Gantenerumab | Double-blind Solanezumab - OLE Gantenerumab | Double-blind Gantenerumab - OLE Gantenerumab
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/18 | 4/27 | 3/28
Other Adverse Events (participants affected / at risk) | 17/18 | 27/27 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo - OLE Gantenerumab (N=18) | Double-blind Solanezumab - OLE Gantenerumab (N=27) | Double-blind Gantenerumab - OLE Gantenerumab (N=28)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo - OLE Gantenerumab (N=18) | Double-blind Solanezumab - OLE Gantenerumab (N=27) | Double-blind Gantenerumab - OLE Gantenerumab (N=28)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (6) | 4 (11)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 2 (4) | 1 (1)
Catheter site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 4 (4) | 5 (6)
Infusion site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 2 (6) | 2 (8) | 5 (6)
Infusion site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site oedema (General disorders) | 1 (2) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion site pruritus (General disorders) | 3 (4) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (3)
Injection site discolouration (General disorders) | 2 (5) | 1 (1) | 3 (3)
Injection site erythema (General disorders) | 8 (97) | 17 (247) | 17 (367)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 2 (5) | 4 (4) | 4 (43)
Injection site mass (General disorders) | 2 (14) | 1 (1) | 1 (21)
Injection site oedema (General disorders) | 0 (0) | 1 (28) | 3 (80)
Injection site pain (General disorders) | 2 (2) | 5 (18) | 9 (28)
Injection site pruritus (General disorders) | 5 (16) | 5 (35) | 8 (88)
Injection site reaction (General disorders) | 1 (1) | 2 (7) | 5 (12)
Injection site swelling (General disorders) | 5 (24) | 7 (100) | 11 (47)
Injection site urticaria (General disorders) | 0 (0) | 1 (2) | 2 (2)
Injection site warmth (General disorders) | 0 (0) | 1 (2) | 2 (5)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 3 (3)
Puncture site erythema (General disorders) | 0 (0) | 0 (0) | 2 (4)
Puncture site pain (General disorders) | 1 (1) | 3 (4) | 4 (4)
Puncture site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 4 (5)
Surgical failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (2) | 3 (3)
Chronic sinusitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (10) | 14 (16) | 15 (17)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (2) | 5 (5)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 5 (9) | 6 (9) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (7) | 2 (3) | 8 (14)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (4)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 3 (3) | 2 (7) | 3 (8)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 (4) | 2 (3) | 3 (3)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (4)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (4)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (5) | 6 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 2 (2) | 5 (7) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 7 (12) | 6 (8) | 5 (9)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Brain stem microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 3 (4) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 3 (3) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Electric shock sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (15) | 8 (20) | 11 (32)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4)
Status migrainosus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 6 (6)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (8) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Menopause (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Pharma Partner and Sponsor decided to terminate the study early based on the status of the drug program and findings from the interim efficacy analysis. The Interim Analysis will be updated here at a later date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's may publish data and study results individually after the earlier of: 1) multi-center Publication is published; 2) no multi-center publication is submitted within 18 months after conclusion, abandonment, or termination of the Protocol at all sites; or 3) sponsor confirms in writing there will be no multi-center Publication. PI must submit results communications to the sponsor at least 75 days prior to submission or presentation. Sponsor can require changes to the communication.

DOCUMENTS (2):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT06424236/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT06424236/SAP_001.pdf